CLINICAL TRIAL: NCT07218666
Title: Phase II Study of Zanzalintinib in Men With Aggressive Variant Prostate Cancer (NAPOLEON Study)
Brief Title: Zanzalintinib in Men With Aggressive Variant Prostate Cancer
Acronym: NAPOLEON
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Deepak Kilari (Other)
Collaborators: Exelixis (Industry); Medical College of Wisconsin (Other)
Responsible Party: Sponsor-Investigator, Deepak Kilari, Sponsor-Investigator, Hoosier Cancer Research Network
Organization: Hoosier Cancer Research Network (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HCRN-GU23-655
Record Dates: First submitted 2025-10-16; First posted 2025-10-20 (Actual); Last update posted 2025-10-21 (Actual); Status verified 2025-10

CONDITIONS: Aggressive Variant Prostate Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Zanzalintinib (Experimental): Zanzalintinib 60mg orally (PO) will be given once daily in subjects with AVPC.
  Interventions: Drug: Zanzalintinib

INTERVENTIONS:
Drug: Zanzalintinib — Zanzalintinib 60mg orally (PO) once daily in
  Other Names: XL092

SUMMARY:
This is a multi-center single arm phase II study to evaluate the antitumor activity of zanzalintinib 60mg orally (PO) once daily in subjects with AVPC. Zanzalintinib may continue until radiographic progression (or beyond), intolerable adverse events, or withdrawal of consent. As long as the subject is clinically stable, subjects may receive study treatment even after radiographic progression, until they are no longer clinically benefiting from the study treatment in the opinion of the treating Investigator, or they need subsequent systemic anticancer treatment or other urgent tumor directed medical intervention to prevent life-threatening complications.

This study will use a 2-stage group-sequential design for enrollment. The first stage will consist of enrolling 15 subjects. No more than 5 of the first 15 subjects can have received chemotherapy in the castrate- resistant setting.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent and HIPAA authorization for release of personal health information prior to registration. NOTE: HIPAA authorization may be included in the informed consent or obtained separately.
2. Age ≥ 18 years at the time of consent.
3. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0-2 within 14 days prior to registration.
4. Histological or cytologically proven prostate cancer
5. Must have had evidence of metastatic disease (AJCC v.8 M1 disease) based on conventional CT/MRI and/or bone scan. This will be defined as:

   * Bone metastases detected by CT, radionuclide 99Tc- methylene bisphosphonate bone scan, or MRI as defined by PCWG3 criteria, OR
   * Non-pelvic lymph node metastases (measurable lymph nodes above the aortic bifurcation; lymph nodes are measurable if the short axis diameter is ≥15 mm) detected on CT or MRI as defined by RECIST version 1.1. Subjects with regional lymph node metastases only (N1, below the aortic bifurcation) will not be eligible for the study; OR
   * Visceral or soft tissue metastases detected on CT or MRI as defined by RECIST version 1.1. Soft tissue/visceral lesions are measurable if the long axis diameter is ≥10 mm.
6. Bilateral orchiectomy or ongoing androgen deprivation therapy with a gonadotropin releasing hormone (GnRH) agonist/antagonist (surgical or medical castration), with serum testosterone < 50 ng/ dL (< 1.73 nmol/L) at screening.
7. Must have progressed during or after at least one second-generation androgen receptor pathway inhibitor (abiraterone acetate, enzalutamide, apalutamide, darolutamide) given for castration-sensitive locally advanced (T3 or T4) or metastatic castration-sensitive prostate cancer (CSPC), M0 castrate- resistant prostate cancer (CRPC), or metastatic CRPC.

   Note: Subjects may have previously received taxane-based chemotherapy for metastatic castration-sensitive prostate cancer (mCSPC), and sipuleucel-T, olaparib, Pluvicto (Lutetium (177Lu) vipivotide tetraxetan), and/or radium-223 for castrate -resistant prostate cancer. The number of patients who have received both taxanes and/or platinum in a CRPC setting will be limited to 5/15 in the first stage and thereby sponsor investigator approval is required prior to enrollment of patients who meet above criteria.
8. Presence of at least one of the following:

   * Presence of visceral metastases or high-volume disease (> 4 sites of metastases) on conventional imaging (CT/MRI/bone scan) with a PSA ≤ 5.
   * Predominantly lytic bone metastasis.
   * Bulky (≥5 cm) lymphadenopathy OR bulky (≥5 cm) high-grade (Gleason ≥8) tumor mass in the prostate/pelvis.
   * Serum chromogranin A level ≥ 5× upper limit of normal (ULN) and/or serum neuron specific enolase (NSE) ≥ 2× ULN.
   * Prostate adenocarcinoma with IHC staining for neuroendocrine markers (positive staining of chromogranin A or synaptophysin).
   * Alterations in at least two of the three tumor suppressor genes: TP53, RB1 and PTEN on genomic testing.
   * Progression to CRPC within 6 months or less of initiation of hormonal therapy.
   * Poorly differentiated or transdifferentiated carcinoma.
   * PSMA negative/FDG avid disease on PET scan.
9. Recovery of adverse events (AEs), including immune-related adverse events (irAEs), to baseline or ≤ Grade 1 severity (CTCAE v5) related to any prior treatments, unless AE(s) are clinically nonsignificant and/or stable on supportive therapy (eg, physiological replacement of corticosteroid). Low-grade or controlled toxicities such as alopecia, ≤ Grade 2 hypomagnesemia, ≤ Grade 2 neuropathy are permitted.
10. Demonstrate adequate organ function as defined in the table below. All screening labs to be obtained within 14 days prior to registration.

    * Platelets (Plt) ≥ 100,000/mm3 without transfusion within 2 weeks of sample collection
    * Absolute Neutrophil Count (ANC) ≥ 1500/mm3 without granulocyte colony-stimulating factor support within 2 weeks of sample collection
    * Hemoglobin (Hgb) ≥ 9 g/dL without transfusion within 2 weeks of sample collection.
    * Calculated creatinine clearance1 ≥ 40 mL/min
    * Urine protein-to-creatinine ratio (UPCR) ≤ 1 mg/mg (≤ 113.2 mg/mmol) creatinine
    * Total bilirubin ≤1.5 × upper limit of normal (ULN); ≤ 3 × ULN for subjects with Gilbert's disease
    * Aspartate aminotransferase (AST) ≤ 3 × ULN
    * Alanine aminotransferase (ALT) ≤ 3 × ULN
    * Alkaline phosphatase (ALP) ≤ 3 × ULN; ≤ 5 × ULN for subjects with documented bone metastasis; ≤ 10 x ULN for subjects with CRPC and bone metastasis if predominantly bone-specific ALP
    * International Normalized Ratio (INR) ≤ 1.5 × ULN
    * Activated Partial Thromboplastin Time (aPTT) ≤ 1.2 × ULN
11. Sexually active fertile subjects and their partners must agree to use highly effective methods of contraception during the course of the study and for 96 days after the last dose of study drug.
12. Projected life expectancy of at least 6 months as determined by treating investigator.
13. Ability of the subject to understand and comply with study procedures for the entire length of the study as determined by the enrolling physician or protocol designee.

Exclusion Criteria:

1. Pure small cell carcinoma of the prostate.
2. Prior treatment with zanzalintinib.
3. Imminent or established spinal cord compression based on clinical and/or imaging findings.
4. Receipt of any type of small molecule kinase inhibitor (including investigational kinase inhibitor) within 2 weeks before first dose of study drug.
5. Receipt of any type of cytotoxic, biologic, or other systemic anticancer therapy (including investigational) within 2 weeks of start of investigational agent and during the study. Concomitant use of megestrol acetate or leuprolide is permitted. The anti-androgen abiraterone is permitted up to 1 week prior to the first dose of study drug. Other types of hormonal therapies with similar use require prior approval of the Sponsor Investigator.
6. Radiation therapy for bone metastasis within 2 weeks or any other radiation therapy within 4 weeks before first dose of study drug. Systemic treatment with radionuclides within 6 weeks before first dose of study drug are not permitted. Subjects with clinically relevant ongoing complications from prior radiation therapy are not eligible.
7. Known brain metastases or cranial epidural disease unless adequately treated with radiotherapy and/or surgery (including radiosurgery) and stable for at least 4 weeks before first dose of study drug. Note: Eligible subjects must be neurologically asymptomatic and without corticosteroid treatment at the time of enrollment. Note: Base of skull lesions without definitive evidence of dural or brain parenchymal involvement are allowed.
8. Concomitant anticoagulation with oral anticoagulants (eg, warfarin, direct thrombin inhibitors) and platelet inhibitors (eg, clopidogrel). Note: Subjects must discontinue prohibited oral anticoagulants within 3 days or 5 half-lives prior to first dose of study drug, whichever is longer.

   The following anticoagulants are allowed:
   1. Prophylactic use of low-dose aspirin for cardio-protection (per local applicable guidelines) and low-dose low molecular weight heparins (LMWH).
   2. Therapeutic doses of LMWH or anticoagulation with direct factor Xa inhibitors rivaroxaban, edoxaban, or apixaban in subjects without known brain metastases who are on a stable dose of the anticoagulant for at least 1 week before first dose of study drug without clinically significant hemorrhagic complications from the anticoagulation regimen.
9. Any complementary medications (eg, herbal supplements or traditional Chinese medicines) to treat the disease under study within 2 weeks before first dose of study drug.
10. The subject has uncontrolled, significant intercurrent or recent illness including, but not limited to, the following conditions:

    a. Unstable deteriorating cardiovascular disorders: i. Congestive heart failure New York Heart Association class 2 or higher, unstable angina pectoris, new-onset angina, serious cardiac arrhythmias (eg, ventricular flutter, ventricular fibrillation, Torsades de pointes).

    ii. Uncontrolled hypertension defined as sustained blood pressure (BP) > 140 mm Hg systolic or > 90 mm Hg diastolic despite optimal antihypertensive treatment.

    iii. Stroke (including transient ischemic attack [TIA]), myocardial infarction, or other clinically significant arterial thrombotic and/or ischemic event within 6 months before first dose of study drug.

    iv. Pulmonary embolism (PE) or deep vein thrombosis (DVT) or prior clinically significant venous events within 3 months before first dose of study drug.

    Note: Subjects with a diagnosis of DVT within 6 months are allowed if asymptomatic and stable at screening and are on a stable dose of the anticoagulant for at least 1 week before first dose of study drug without clinically significant hemorrhagic complications from the anticoagulation regimen.

    Note: Subjects who don't require prior anticoagulation therapy may be eligible but must be discussed and approved by the Sponsor Investigator.

    b. Gastrointestinal (GI) disorders including those associated with a high risk of perforation or fistula formation: i. Tumors invading the GI-tract from external viscera. ii. Active peptic ulcer disease, inflammatory bowel disease, diverticulitis, cholecystitis, symptomatic cholangitis or appendicitis, or acute pancreatitis iii. Acute obstruction of the bowel, gastric outlet, or pancreatic or biliary duct within 6 months before first dose unless cause of obstruction is definitively managed and subject is asymptomatic.

    iv. Abdominal fistula, gastrointestinal perforation, bowel obstruction, or intra-abdominal abscess within 6 months before first dose. Note: Complete healing of an intra-abdominal abscess must be confirmed before first dose of study drug.

    v. Known gastric or esophageal varices. vi. Ascites, pleural effusion, or pericardial fluid requiring drainage in last 4 weeks before first dose of study drug.
11. Clinically significant hematuria, hematemesis, or hemoptysis of > 0.5 teaspoon (2.5 ml) of red blood, or other history of significant bleeding (eg, pulmonary hemorrhage) within 12 weeks before first dose of study drug.
12. Symptomatic cavitating pulmonary lesion(s) or endobronchial disease (asymptomatic or radiated lesions allowed)
13. Lesions invading major blood vessel including, but not limited to, inferior vena cava, pulmonary artery, or aorta. Note: Subjects with intravascular tumor extension (eg, tumor thrombus in renal vein or inferior V. cava) may be eligible following Sponsor Investigator approval.
14. Other clinically significant disorders that would preclude safe study participation.

    a Active infection requiring systemic treatment. Note: Prophylactic antimicrobial treatments (antibiotics, antimycotic, antiviral) are allowed.

    b Known infection with acute or chronic hepatitis B or C. Note: Hepatitis B and C testing will be performed at screening.

    c Known human immunodeficiency virus (HIV) or acquired immunodeficiency syndrome (AIDS)-related illness except for subjects meeting all of the following criteria: i. on stable anti-retroviral therapy, and ii. CD4+ T cell count ≥ 200/µL, and iii. an undetectable viral load. Note: HIV testing will be performed at screening if and as required by local regulation.

    Note: To be eligible, participants taking CYP inhibitors (eg, zidovudine, ritonavir, cobicistat, didanosine) or CYP3 inducers (efavirenz) must change to a different regimen not including these drugs 7 days prior to initiation of study treatment. Anti-retroviral therapies (ART) must have been received for at least 4 weeks prior to the first dose.

    Note: CD4+ T cell counts, and viral load are monitored per standard of care by the local health care provider.

    c Serious non-healing wound/ulcer/bone fracture. Note: non-healing wounds or ulcers are permitted if due to tumor-associated skin lesions.

    d Malabsorption syndrome e Pharmacologically uncompensated, symptomatic hypothyroidism f Moderate to severe hepatic impairment (Child-Pugh B or C) g Requirement for hemodialysis or peritoneal dialysis. h History of solid organ or allogeneic stem cell transplant.
15. Major surgery (as defined in Section 5.2.5; eg, GI surgery, removal or biopsy of brain metastasis) within 8 weeks prior to first dose of study treatment. Prior laparoscopic surgeries (ie nephrectomy) within 4 weeks prior to first dose of study treatment. Minor surgery (eg, simple excision, tooth extraction) within 5 days before first dose of study treatment. Complete wound healing from major or minor surgery must have occurred at least prior to first dose of study drug. Note: Fresh tumor biopsies should be performed at least 5 days before the first dose of study treatment. Subjects with clinically relevant ongoing complications from prior surgical procedures, including biopsies, are not eligible.
16. Corrected QT interval calculated by the Fridericia formula (QTcF) > 480 ms per electrocardiogram (ECG) performed within 14 days before first dose of study treatment. Note: Triplicate ECG evaluations will be performed and the average of these 3 consecutive results for QTcF will be used to determine eligibility.
17. History of psychiatric illness likely to interfere with ability to comply with protocol requirements or give informed consent.
18. Inability to swallow tablets or ingest a suspension either orally or by a nasogastric (NG) or gastrostomy (PEG) tube.
19. Previously identified allergy or hypersensitivity to components of the study treatment formulations.
20. Prior malignancy which required active therapy within 2 years before first dose of study drug.

    Notes:
    * Inclusion of patients with prior malignancies is allowed if the risk of the prior malignancy interfering with either safety or efficacy end points is very low, as assessed by the treating investigator.
    * Patients with a previously treated malignancy are eligible to participate if all treatment of that malignancy was completed at least 2 years before registration and the patient has no evidence of disease.
    * Patients who have a concurrent malignancy that is clinically stable and does not require tumor-directed treatment are allowed to participate.
21. Other conditions which, in the opinion of the treating Investigator, would compromise the safety of the patient or the patient's ability to complete the study.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-05 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Radiographic progression free survival (rPFS) | 6 months
  For soft tissue lesions, rPFS is defined as the date of Cycle 1 Day 1 to date of radiologic progression of soft tissue lesions per RECIST 1.1 or death whichever occurs first.
Radiographic progression free survival (rPFS) | 6 months
  For bone lesions, rPFS is defined as the date of Cycle 1 Day 1 to date of progression of bone lesions per PCWG3 criteria or death whichever occurs first.

SECONDARY OUTCOMES:
Adverse Events | 4 years
  Safety of the zanzalintinib will be assessed based on Common Terminology Criteria for Adverse Events (CTCAE) version 5.0
Overall Survival | 4 years
  Overall survival (OS) will be measured from date of registration to date of death from any cause censored at the date of last follow-up.
Objective response rate (ORR) | 4 years
  ORR will be the proportion of patients with measurable disease achieving either a confirmed complete response or a partial response per RECIST 1.1 for patients with measurable disease.
Duration of response (DoR) | 4 years
  DOR will be measured from the time a partial response or complete response is first noted until the date of progression as defined by RECIST version 1.1 for patients with measurable disease.
Quality of life (QOL) | 4 years
  QOL will be assessed by changes in FACT-P. The response scale is a 5-point Likert-type scale with 0 being the minimum value and 4 being the maximum value for each individual question. The minimum score for the entire questionnaire is 0 and the maximum score is 156. The higher the score, the better the quality of life.
Time to first subsequent anti-cancer therapy or death | 4 years
  Time to first subsequent anti-cancer treatment will be defined as the time from the start of a zanzalintinib to the start of the next line of therapy or death. Subjects alive without a next line of therapy at the end of follow-up will be censored.

CONTACTS AND LOCATIONS:
Overall Officials: Deepak Kilari, MD, Principal Investigator — Medical College of Wisconsin